CLINICAL TRIAL: NCT00015301
Title: Methylphenidate Raclopride PET Test
Brief Title: Methylphenidate Raclopride Positron Emission Tomography (PET) Test - 11
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: New York MDRU (Other)
Masking: Double | Purpose: Diagnostic
Other Study IDs: NIDA-5-0013-11; Y01-5-0013-11
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Methylphenidate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Methylphenidate

SUMMARY:
The purpose of this study is to evaluate PET methodology to study in vivo synaptic dopamine release.

DETAILED DESCRIPTION:
The objective of this study is to evaluate PET methodology to study in vivo synaptic dopamine release.

ELIGIBILITY:
Inclusion Criteria:

Healthy normals

Exclusion Criteria:

History of head trauma or loss of consciousness. Significant medical history. History of seizures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 2003-12 (Actual); Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Dopamine receptor availability

CONTACTS AND LOCATIONS:
Overall Officials: John Rotrosen, M.D., Principal Investigator — New York MDRU
Locations (1):
- New York MDRU, New York, New York, United States